CLINICAL TRIAL: NCT04775667
Title: Kinesiophobia and Associated Factors in Patients With Traumatic Lower Extremity Amputation
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Physical Medicine and Rehabilitation Associate Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 12
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Amputation
Keywords: kinesiophobia; amputation; pain; fear of fall; quality of life
MeSH Terms: conditions — Kinesiophobia; Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaires for clinical assessments — questionnaires for clinical assessments

SUMMARY:
There are limited studies examining kinesiophobia and factors associated with kinesophobia in patients with lower limb amputation. The aim of this study is to illustrate the level of kinesiophobia in patients with traumatic lower extremity amputation and to analyze the correlation between kinesiophobia and associated factors (pain, prosthesis satisfaction, fear of fall, quality of life). This cross-sectional study will involve 52 patients with traumatic lower extremity amputation. Kinesiophobia level will be measured with the Tampa Scale for Kinesiophobia (TSK). All patients will point the severity of sound limb pain, residual limb pain, low back pain and the overall prosthesis, socket system and prosthetic foot satisfaction on a Visual Analogue Scale (VAS). Falls Efficacy Scale-International (FES-I) will be used for evaluation of falls efficacy under different circumstances. The quality of life (QoL) will be assessed with Nottingham Health Profile (NHP).

DETAILED DESCRIPTION:
Kinesiophobia is defined as an unreasonable, excessive, and debilitating fear of physical activity and movement resulting from a feeling of susceptibility to painful injury or re-injury. Kinesiophobia was demonstrated to be related to lower levels of physical activity in people with chronic pain. As a result, there is an increased risk of sedentary lifestyle. Inactivity increases the risk of chronic pain as well as other health problems such as cardiovascular diseases. Kinesiophobia also is related to poor treatment outcomes. The negative effects of kinesiophobia on rehabilitation processes including exercise programs and thus its importance in the clinical course were illustrated in studies on various diseases.

There are limited studies examining kinesiophobia and factors associated with kinesophobia in patients with lower limb amputation. The aim of this study is to illustrate the level of kinesiophobia in patients with traumatic lower extremity amputation and to analyze the correlation between kinesiophobia and associated factors (pain, prosthesis satisfaction, fear of fall, quality of life).

his cross-sectional study will involve 52 patients with traumatic lower extremity amputation. Kinesiophobia level will be measured with the Tampa Scale for Kinesiophobia (TSK). All patients will point the severity of sound limb pain, residual limb pain, low back pain and the overall prosthesis, socket system and prosthetic foot satisfaction on a Visual Analogue Scale (VAS). Falls Efficacy Scale-International (FES-I) will be used for evaluation of falls efficacy under different circumstances. The quality of life (QoL) will be assessed with Nottingham Health Profile (NHP).

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-65 years
2. time after amputation ≥ 6 months
3. unilateral or bilateral amputation above the ankle level
4. using a prosthesis

Exclusion Criteria:

1. upper extremity amputation
2. the presence of musculoskeletal or neurological disease that could cause functional impairment other than amputation
3. the presence of neurological deficit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with traumatic lower extremity amputation
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Tampa Scale for Kinesiophobia (TSK) | through study completion, an average of one and a half months
  Kinesiophobia level will be measured with the Tampa Scale for Kinesiophobia (TSK). The questionnaire contains 17 items that uses a 4-point Likert-type scale (from 1 (strongly disagree) to 4 (strongly agree)). A score of 39 or above will be used in order to distinguish those with a high level of kinesophobia. The validity and reliability of the Turkish version of TKS has been demonstrated.
Visual Analogue Scale (VAS) | through study completion, an average of one and a half months
  All patients will point the severity of sound limb pain, residual limb pain, low back pain and the overall prosthesis, socket system and prosthetic foot satisfaction on a Visua Analogue Scale (VAS; from 0 (no pain) to 10 (worst pain)).
Falls Efficacy Scale-International (FES-I) | through study completion, an average of one and a half months
  Falls Efficacy Scale-International (FES-I) will be used for evaluation of falls efficacy under different circumstances. The FES-I is a self-report questionnaire, containing 16 items scored on a four-point scale (from 1 (no fear whatsoever) to 4 (very fearful)). The questionnaire provides information about the level of concern associated with falls during 16 various activities of daily living.
Nottingham Health Profile (NHP) | through study completion, an average of one and a half months
  The quality of life (QoL) will be assessed with Nottingham Health Profile (NHP). NHP consists of 38 questions on six different subscales that include physical activity, pain, sleep, fatigue, social isolation and emotional reactions. Each subscale of NHP is scored between 0 and 100, and higher scores illustrate a decrease in QoL. It has been shown that NHP is a reliable scale for measuring health-related quality of life in patients with amputation.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Orucu Atar, Principal Investigator — Gaziler Physical Medicine and Rehabilitation, Training and Research Hospital, Department of PMR
Locations (1):
- Gaziler Physical Medicine and Rehabilitation, Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No